CLINICAL TRIAL: NCT07110610
Title: A First-in-Human, Randomized, Double-Blind, Placebo-Controlled, Phase 1, Single and Multiple Ascending Dose Study of LTG-321 Administered Orally to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Healthy Male and Female Participants 18 to 55 Years of Age
Brief Title: Phase 1 Single and Multiple Ascending Dose of LTG-321 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Latigo Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTG-321-013
Record Dates: First submitted 2025-07-01; First posted 2025-08-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTG-321 (Experimental): receives active investigational drug
  Interventions: Drug: LTG-321
- Placebo (Placebo Comparator): receives placebo comparator
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LTG-321 — active investigational drug
  Arms: LTG-321
Other: Placebo — Placebo-to-match LTG-321
  Arms: Placebo

SUMMARY:
This is a first-in-human, randomized, double-blind, placebo-controlled Phase 1 single ascending dose (SAD) and multiple ascending dose (MAD) study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of orally administered LTG-321 in healthy male and female participants 18 to 55 years of age. The study will be conducted in New Zealand.

The study also includes a randomized, double-blind, placebo-controlled, within-participant crossover evaluation of pain tolerance using a cold pressor test in healthy male participants 18 to 55 years of age. In addition, a randomized, open-label, crossover Food Effect cohort will evaluate the impact of a high-fat meal on the pharmacokinetics of LTG-321 following single oral doses in the fed and fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 to 55 years, inclusive, at the time of signing the informed consent.
* Overtly healthy with no clinically relevant abnormalities based on the medical history, physical examinations, clinical laboratory evaluations, and 12-lead ECG that, in the opinion of the investigator, would affect participant safety.
* Body mass index (BMI) within the range of 18-30 kg/m2 (inclusive).

Exclusion Criteria:

* Inability to take oral medications or gastrointestinal abnormalities potentially impacting absorption.
* Clinically significant cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, gastrointestinal, immunological, dermatological, neurological, or psychiatric disease which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the investigator, unacceptably increase the participant's risk by participating in the study.
* Past or current history or evidence of alcohol abuse and/or dependence on recreational drug use
* Donation of over 500 mL blood ≤ 3 months prior to start of participation
* Participant is under legal custodianship.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the Incidence, severity, seriousness, and causality of treatment-emergent adverse events (TEAEs) of single and multiple ascending oral doses of LTG-321 in healthy participants | Up to 14 days of dosing
  Incidence, severity, seriousness, and causality of treatment-emergent adverse events (TEAEs)
To evaluate the Pain Detection and Tolerance Threshold during Cold Pressor Test of LTG-321 in healthy male participants. | Up to 5 days of dosing
  Change from baseline at various individual time points and at various intervals for time to reach pain detection threshold (PDT) and time to reach pain tolerance threshold (PTT), for each dose of LTG-321 vs. placebo.
Effect of Food on Pharmacokinetics of LTG-321 | Up to approximately 48 hours post-dose in each treatment period
  Assessment of the effect of a high-fat meal on systemic exposure of LTG-321 following a single oral dose administered under fed and fasted conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No